CLINICAL TRIAL: NCT06926673
Title: A Phase II, Randomized, Open-label Platform Trial Utilizing a Master Protocol to Study Novel Regimens Versus Standard of Care Treatment in NSCLC Participants
Brief Title: Platform Trial of Novel Regimens Versus Standard of Care (SoC) in Participants With Non-small Cell Lung Cancer (NSCLC) - Sub-study 3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 205801-003; 2018-001316-29 (EudraCT Number)
Record Dates: First submitted 2025-04-11; First posted 2025-04-14 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms
Keywords: NSCLC; Dostarlimab; Belrestotug; Nelistotug
MeSH Terms: conditions — Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dostarlimab plus Belrestotug (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Belrestotug.
- Dostarlimab plus Belrestotug plus Nelistotug (Experimental)
  Interventions: Drug: Dostarlimab; Drug: Belrestotug.; Drug: Nelistotug

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab will be administered
Drug: Belrestotug. — Belrestotug will be administered
Drug: Nelistotug — Nelistotug will be administered.
  Arms: Dostarlimab plus Belrestotug plus Nelistotug

SUMMARY:
This study is a sub-study of the master protocol 205801 (NCT03739710). This sub study will assess safety and pharmacokinetics and pharmacodynamics (PK/PD) of novel regimens (Dostarlimab plus belrestotug , and Dostarlimab plus belrestotug plus nelistotug) in participants with previously treated NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of giving signed informed consent/assent.
* Male or female, aged 18 years or older at the time consent is obtained.
* Participants with histologically or cytologically confirmed diagnosis of NSCLC (squamous or non-squamous) and

  1. Documented disease progression based on radiographic imaging, during or after a maximum of 2 lines of systemic treatment for locally/regionally advanced recurrent, Stage IIIb/Stage IIIc/Stage IV or metastatic disease. Two components of treatment must have been received in the same line or as separate lines of therapy: i) No more than or less than 1 line of platinum-containing chemotherapy regimen, and ii) No more than or less than 1 line of Programmed cell death ligand 1 (PD[L]1) monoclonal antibody (mAb) containing regimen.
  2. Participants with known V-Raf Murine Sarcoma Viral Oncogene Homolog B (BRAF) molecular alterations must have had disease progression after receiving the locally available SoC treatment for the molecular alteration.
  3. Participants who received prior anti-PD(L)1 therapy must fulfill the following requirements: i) Have achieved a CR, PR or SD and subsequently had disease progression (per RECIST 1.1 criteria) either on or after completing PD(L)1 therapy ii) Have not progressed or recurred within the first 12 weeks of PD(L)1 therapy, either clinically or per RECIST 1.1 criteria
* Measurable disease, presenting with at least 1 measurable lesion per RECIST 1.1.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1.
* A tumor tissue sample obtained at any time from the initial diagnosis of NSCLC to time of study entry is mandatory. Although a fresh tumor tissue sample obtained during screening is preferred, archival tumor specimen is acceptable.
* Adequate organ function as defined in the protocol.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least 1 of the following conditions apply:

  i) Not a woman of childbearing potential (WOCBP) as defined in the protocol or ii) A WOCBP who agrees to follow the protocol defined contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* Life expectancy of at least 12 weeks.

Exclusion Criteria:

Participants who received prior treatment with the following therapies (calculation is based on date of last therapy to date of first dose of study treatment):

1. Docetaxel at any time.
2. Any of the investigational agents being tested in the current study.
3. Systemic approved or investigational anticancer therapy within 30 days or 5 half-lives of the drug, whichever is shorter. At least 14 days must have elapsed between the last dose of prior anticancer agent and the first dose of study drug administered.
4. Prior radiation therapy: permissible if at least one non-irradiated measurable lesion is available for assessment per RECIST version 1.1 or if a solitary measurable lesion was irradiated, objective progression is documented. A wash out of at least 2 weeks before start of study drug for radiation of any intended use is required.

   * Received greater than (>) 2 prior lines of therapy for NSCLC, including participants with BRAF molecular alternations.
   * Invasive malignancy or history of invasive malignancy other than disease under study within the last 2 years.
   * Carcinomatous meningitis (regardless of clinical status) and uncontrolled or symptomatic Central nervous system (CNS) metastases.
   * Major surgery less than or equal to (<=) 28 days of first dose of study treatment.
   * Autoimmune disease (current or history) or syndrome that required systemic treatment within the past 2 years. Replacement therapies which include physiological doses of corticosteroids for treatment of endocrinopathies (for example, adrenal insufficiency) are not considered systemic treatments.
   * Receiving systemic steroids (>10 milligrams [mg]) oral prednisone or equivalent) or other immunosuppressive agents within 7 days prior to first dose of study treatment. Steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication) are permitted.
   * Prior allogeneic/autologous bone marrow or solid organ transplantation.
   * Receipt of any live vaccine within 30 days prior to first dose of study treatment.
   * Toxicity from previous anticancer treatment that includes:

1. Greater than or equal to (>=) Grade 3 toxicity considered related to prior immunotherapy and that led to treatment discontinuation.

2. History of myocarditis of any grade during a previous treatment with immunotherapy 3. Toxicity related to prior treatment that has not resolved to <= Grade 1 (except alopecia, hearing loss, endocrinopathy managed with replacement therapy, and peripheral neuropathy which must be <= Grade 2).

* History (current and past) of idiopathic pulmonary fibrosis, pneumonitis (for pastpneumonitis exclusion only if steroids were required for treatment), interstitial lung disease, or organizing pneumonia.
* Recent history (within the past 6 months) of uncontrolled symptomatic ascites, pleural or pericardial effusions.
* Recent history (within the past 6 months) of gastrointestinal obstruction that required surgery, acute diverticulitis, inflammatory bowel disease, or intra-abdominal abscess.
* History or evidence of cardiac abnormalities within the 6 months prior to enrollment which include

  1. Serious, uncontrolled cardiac arrhythmia or clinically significant electrocardiogram abnormalities including second degree (Type II) or third degree atrioventricular block.
  2. Cardiomyopathy, myocardial infarction, acute coronary syndromes (including unstable angina pectoris), coronary angioplasty, stenting or bypass grafting.
  3. Symptomatic pericarditis.
* Current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypo-albuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Active infection requiring systemic therapy <=7 days prior to first dose of study treatment.
* Participants with known human immunodeficiency virus infection.
* Participants with history of severe hypersensitivity to mAbs or hypersensitivity to any of the study treatment(s) or their excipients.
* Any serious and/or unstable pre-existing medical (aside from malignancy), psychiatric disorder, or other condition that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures in the opinion of the investigator.
* Pregnant or lactating female participants.
* Participant who is currently participating in or has participated in a study of an investigational device within 4 weeks prior to the first dose of study treatment.
* Participants with presence of hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Participants with positive hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study treatment.
* Receipt of transfusion of blood products (including platelets or red blood cells) or administration of colony-stimulating factors (including granulocyte colony stimulating factor [G-CSF], granulocyte-macrophage colony-stimulating factor, and recombinant erythropoietin) within 14 days before the first dose of study intervention.
* Known hypersensitivity to components or excipients of dostarlimab, belrestotug, and/or nelistotug
* Has received prior antibodies or drugs targeting TIGIT, CD96, PVRIG, or other therapies targeting the CD226 axis pathway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- GSK Investigational SIte, Nashville, Tennessee, United States
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Toronto, Ontario
- France (3):
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Großhansdorf, Germany
- Italy (3):
  - GSK Investigational Site, Meldola FC
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Siena
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga

IPD SHARING:
Plan to Share IPD: Yes
Study Sponsor will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a sub-study of the master study NCT03739710.The master protocol included two parts -Part 1 (non-randomized, safety and PK/PD evaluation) and Part 2 (randomized part comparing safety and efficacy to SoC). Criteria on whether to advance a study regimen from Part 1 to Part 2 has been built into the study design. Having completed Part 1 with the allowable number of patients per protocol, the decision was taken to not enroll participants in Part 2. Part 1 was therefore considered completed.
Groups:
- Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)]: Participants with Non-Small Cell Lung Cancer (NSCLC) were administered with 500 milligrams (mg) of Dostarlimab as IV infusion once every 3 weeks (Q3W) in combination with Belrestotug LD as IV infusion Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met.
- Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)]: Participants with NSCLC were administered with 500 mg of Dostarlimab as IV infusion Q3W in combination with Belrestotug MD as IV infusion Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met.
- Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]: Participants with NSCLC were administered with 500 mg of Dostarlimab as IV infusion once Q3W in combination with Belrestotug HD as IV infusion Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met.
- Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD: Participants with NSCLC received 500 mg Dostarlimab followed by Belrestotug MD and Nelistotug MD. Treatment were given via IV infusion from day 1 to Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met. Participants in this safety part were evaluated to determine the maximum tolerable dose tested.
- Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD: Participants with NSCLC received 500 mg Dostarlimab followed by Belrestotug MD and Nelistotug HD. Treatment were given via IV infusion from day 1 to Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met. Participants in this safety part were evaluated to determine the maximum tolerable dose tested.
- Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD: Participants with NSCLC received 500 mg Dostarlimab followed by Belrestotug MD and Nelistotug LD. Treatment were given via IV infusion from day 1 to Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met. In this randomization part, participants were assessed for pharmacokinetics/pharmacodynamics (PK/PD) and received Nelistotug LD
- Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD: Participants with NSCLC received 500 mg Dostarlimab followed by Belrestotug MD and Nelistotug HD. Treatment were given via IV infusion from day 1 to Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met. In this randomization part, participants were assessed for PK/PD and received Nelistotug HD.
Period: Overall Study
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Started (Enrolled Set Population included all participants who passed screening and were assigned treatment.) | 6 | 9 | 9 | 10 | 7 | 11 | 10
DLT Evaluable Population (All participants who took at least one dose of study treatment and followed for the DLT observation period or were withdrew within the DLT observation period due to meeting the DLT criteria and no resolution/recovery.) | 0 | 4 | 4 | 4 | 7 | 0 | 0
Completed (Participants who completed follow-up or who died were considered to have completed the study.) | 6 (2 participants completed follow-up and 4 died) | 6 (1 participant completed follow-up and 5 died) | 7 (7 participants died) | 8 (1 participant completed follow-up and 7 died) | 7 (3 participants completed follow-up and 4 died) | 9 (2 participant completed follow-up and 7 died) | 9 (3 participants completed follow-up and 6 died)
Not Completed | 0 | 3 | 2 | 2 | 0 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 2 | 1 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Total
Number analyzed (Participants) | 6 | 9 | 9 | 10 | 7 | 11 | 10 | 62
Age, Customized [Count of Participants; unit: Participants]
  18 to >=85 years | 6 | 9 | 9 | 10 | 7 | 11 | 10 | 62
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 5 | 3 | 4 | 4 | 26
  Male | 3 | 6 | 5 | 5 | 4 | 7 | 6 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 7 | 8 | 10 | 6 | 8 | 5 | 48
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 1 | 0 | 0 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Any Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) (Arm 4)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose resulted in death, is life threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/ incapacity, is a congenital anomaly/ birth defect, other situations and is associated with liver injury or impaired liver function. SAEs are subset of AEs. A TEAE is any event that was not present prior to the initiation of study treatment or any event already present that worsens in either intensity or frequency following exposure to study treatment. AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA) coding system.
Time Frame: Up to approximately 97 weeks
Population: Safety Population included all participants who received at least 1 dose of standard of care (SoC) or experimental regimen based on actual treatment received.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 9
Participants
  Any TEAEs | 6 | 9 | 8
  Any SAEs | 0 | 3 | 2

2. Primary Outcome: Part 1: Number of Participants With Any TEAEs and SAEs (Arm 5)
Description: as for outcome 1
Time Frame: Up to approximately 107 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants
  Any TEAEs | 10 | 6 | 11 | 9
  Any SAEs | 3 | 3 | 3 | 3

3. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicity (DLT) (Arm 4 and Arm 5)
Description: A DLT is an AE meeting criteria such as, hematologic toxicities of Grade (G) 4 neutropenia/anemia/thrombocytopenia (G3 if bleeding). Non-hematological toxicities include persistent G2 eye events, colitis/diarrhea (G2 unresolved to ≤ G1 within 7 days despite immunosuppressive therapy, G3 for ≥ 72 hours, any G4), G3 pneumonitis, rash (unresolved to ≤ G2 within 2 weeks despite treatment), hypersensitivity/IRR, liver events meeting Hy's Law criteria. G3 toxicity unresolved to ≤G1 or baseline within 3 days with supportive care, or any G4 toxicity. Exclusions include G3 events of electrolyte imbalances correctable within 72 hours without effects, nausea/vomiting/fatigue resolving within 7 days, lymphopenia, and enzyme elevations without pancreatitis. Considerations for DLTs include permanent treatment discontinuation, investigator/sponsor judgment-based events including post-observation period toxicities.
Time Frame: Up to 21 days
Population: DLT-evaluable participants included all participants who took at least 1 dose of study intervention and were followed for the DLT observation period or were withdrawn within the DLT observation period due to meeting the DLT criteria and no resolution/recovery per dose modifications and toxicity management guidelines.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 4 | 4 | 4 | 7
Participants | 0 | 0 | 0 | 1

4. Primary Outcome: Part 1: Number of Participants Requiring Dose Modifications (Arm 4)
Description: Number of participants with dose modifications (missed doses, dose delays and infusion interruptions) is summarized.
Time Frame: Up to approximately 97 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 9
Participants
  Missed Doses | 0 | 3 | 2
  Dose Delays | 0 | 1 | 1
  Infusion Interruptions | 0 | 1 | 1

5. Primary Outcome: Part 1: Number of Participants Requiring Dose Modifications (Arm 5)
Description: Number of participants with dose modifications (missed doses, dose delays and infusion interruptions) is summarized.
Time Frame: Up to approximately 107 weeks
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants
  Missed Doses | 6 | 2 | 5 | 6
  Dose Delays | 1 | 0 | 0 | 0
  Infusion Interruptions | 0 | 2 | 0 | 0

6. Primary Outcome: Part 1: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (Arm 4)
Description: Performance Status was assessed using the ECOG scale (Grades 0-5), where 0: Fully active, able to carry on all pre-disease performance without restriction. Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of light or sedentary nature; Grade 2 - Ambulatory & capable of all self-care but unable to carry out any work activities. Up and about more than (>) 50% of waking hours; Grade 3 -Capable of only limited self-care, confined to bed or chair > 50% of waking hours; Grade 4 -Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; Grade 5 -Dead.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 9
Participants
  Baseline, Grade 0 | 0 | 5 | 3
  Baseline, Grade 1 | 6 | 4 | 6
  Week 4, Grade 0: number analyzed (Participants) | 6 | 8 | 8
  Week 4, Grade 0 | 1 | 4 | 3
  Week 4, Grade 1: number analyzed (Participants) | 6 | 8 | 8
  Week 4, Grade 1 | 3 | 3 | 4
  Week 4, Grade 2: number analyzed (Participants) | 6 | 8 | 8
  Week 4, Grade 2 | 2 | 1 | 1
  Week 7, Grade 0: number analyzed (Participants) | 2 | 3 | 6
  Week 7, Grade 0 | 1 | 2 | 1
  Week 7, Grade 1: number analyzed (Participants) | 2 | 3 | 6
  Week 7, Grade 1 | 1 | 1 | 5
  Week 10, Grade 0: number analyzed (Participants) | 1 | 3 | 4
  Week 10, Grade 0 | 1 | 2 | 1
  Week 10, Grade 1: number analyzed (Participants) | 1 | 3 | 4
  Week 10, Grade 1 | 0 | 1 | 3
  Week 13, Grade 0: number analyzed (Participants) | 1 | 3 | 2
  Week 13, Grade 0 | 1 | 1 | 1
  Week 13, Grade 1: number analyzed (Participants) | 1 | 3 | 2
  Week 13, Grade 1 | 0 | 2 | 1
  Week 16, Grade 0: number analyzed (Participants) | 1 | 3 | 1
  Week 16, Grade 0 | 1 | 1 | 1
  Week 16, Grade 1: number analyzed (Participants) | 1 | 3 | 1
  Week 16, Grade 1 | 0 | 2 | 0
  Week 19, Grade 0: number analyzed (Participants) | 1 | 3 | 1
  Week 19, Grade 0 | 1 | 0 | 1
  Week 19, Grade 1: number analyzed (Participants) | 1 | 3 | 1
  Week 19, Grade 1 | 0 | 3 | 0
  Week 22, Grade 0: number analyzed (Participants) | 1 | 2 | 1
  Week 22, Grade 0 | 1 | 0 | 0
  Week 22, Grade 1: number analyzed (Participants) | 1 | 2 | 1
  Week 22, Grade 1 | 0 | 2 | 1
  Week 25, Grade 0: number analyzed (Participants) | 0 | 2 | 1
  Week 25, Grade 0 |  | 1 | 0
  Week 25, Grade 1: number analyzed (Participants) | 0 | 2 | 1
  Week 25, Grade 1 |  | 1 | 1
  Week 28, Grade 0: number analyzed (Participants) | 0 | 2 | 1
  Week 28, Grade 0 |  | 1 | 0
  Week 28 Grade 1: number analyzed (Participants) | 0 | 2 | 1
  Week 28 Grade 1 |  | 1 | 1
  Week 31, Grade 0: number analyzed (Participants) | 0 | 1 | 1
  Week 31, Grade 0 |  | 1 | 1
  Week 34, Grade 0: number analyzed (Participants) | 0 | 0 | 1
  Week 34, Grade 0 |  |  | 1
  Week 37, Grade 0: number analyzed (Participants) | 0 | 1 | 1
  Week 37, Grade 0 |  | 1 | 1
  Week 40, Grade 0: number analyzed (Participants) | 0 | 1 | 0
  Week 40, Grade 0 |  | 1 |
  Week 43, Grade 0: number analyzed (Participants) | 0 | 1 | 0
  Week 43, Grade 0 |  | 1 |
  Week 46, Grade 0: number analyzed (Participants) | 0 | 1 | 0
  Week 46, Grade 0 |  | 1 |
  Week 49, Grade 0: number analyzed (Participants) | 0 | 1 | 0
  Week 49, Grade 0 |  | 1 |
  Week 52, Grade 1: number analyzed (Participants) | 0 | 1 | 0
  Week 52, Grade 1 |  | 1 |
  Week 55, Grade 1: number analyzed (Participants) | 0 | 1 | 0
  Week 55, Grade 1 |  | 1 |
  Week 58, Grade 0: number analyzed (Participants) | 0 | 1 | 0
  Week 58, Grade 0 |  | 1 |
  Week 61, Grade 0: number analyzed (Participants) | 0 | 1 | 0
  Week 61, Grade 0 |  | 1 |
  Week 64, Grade 1: number analyzed (Participants) | 0 | 1 | 0
  Week 64, Grade 1 |  | 1 |
  Week 67, Grade 1: number analyzed (Participants) | 0 | 1 | 0
  Week 67, Grade 1 |  | 1 |
  Week 70, Grade 1: number analyzed (Participants) | 0 | 1 | 0
  Week 70, Grade 1 |  | 1 |
  Treatment Discontinuation (up to 97 weeks), Grade 0: number analyzed (Participants) | 6 | 7 | 6
  Treatment Discontinuation (up to 97 weeks), Grade 0 | 1 | 1 | 0
  Treatment Discontinuation (up to 97 weeks), Grade 1: number analyzed (Participants) | 6 | 7 | 6
  Treatment Discontinuation (up to 97 weeks), Grade 1 | 2 | 5 | 4
  Treatment Discontinuation (up to 97 weeks), Grade 2: number analyzed (Participants) | 6 | 7 | 6
  Treatment Discontinuation (up to 97 weeks), Grade 2 | 1 | 1 | 1
  Treatment Discontinuation (up to 97 weeks), Grade 3: number analyzed (Participants) | 6 | 7 | 6
  Treatment Discontinuation (up to 97 weeks), Grade 3 | 2 | 0 | 1

7. Primary Outcome: Part 1: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status (Arm 5)
Description: as for outcome 6
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants
  Baseline, Grade 0 | 4 | 2 | 7 | 1
  Baseline, Grade 1 | 6 | 5 | 4 | 9
  Week 4, Grade 0: number analyzed (Participants) | 10 | 6 | 11 | 9
  Week 4, Grade 0 | 4 | 1 | 5 | 1
  Week 4, Grade 1: number analyzed (Participants) | 10 | 6 | 11 | 9
  Week 4, Grade 1 | 4 | 5 | 6 | 8
  Week 4, Grade 2: number analyzed (Participants) | 10 | 6 | 11 | 9
  Week 4, Grade 2 | 2 | 0 | 0 | 0
  Week 7, Grade 0: number analyzed (Participants) | 8 | 4 | 8 | 7
  Week 7, Grade 0 | 3 | 2 | 3 | 1
  Week 7, Grade 1: number analyzed (Participants) | 8 | 4 | 8 | 7
  Week 7, Grade 1 | 3 | 2 | 4 | 6
  Week 7, Grade 2: number analyzed (Participants) | 8 | 4 | 8 | 7
  Week 7, Grade 2 | 2 | 0 | 1 | 0
  Week 10, Grade 0: number analyzed (Participants) | 7 | 3 | 6 | 4
  Week 10, Grade 0 | 1 | 2 | 3 | 1
  Week 10, Grade 1: number analyzed (Participants) | 7 | 3 | 6 | 4
  Week 10, Grade 1 | 5 | 1 | 3 | 3
  Week 10, Grade 2: number analyzed (Participants) | 7 | 3 | 6 | 4
  Week 10, Grade 2 | 1 | 0 | 0 | 0
  Week 13, Grade 0: number analyzed (Participants) | 5 | 2 | 4 | 4
  Week 13, Grade 0 | 2 | 2 | 2 | 0
  Week 13, Grade 1: number analyzed (Participants) | 5 | 2 | 4 | 4
  Week 13, Grade 1 | 3 | 0 | 2 | 4
  Week 16, Grade 0: number analyzed (Participants) | 4 | 2 | 4 | 3
  Week 16, Grade 0 | 2 | 2 | 2 | 1
  Week 16, Grade 1: number analyzed (Participants) | 4 | 2 | 4 | 3
  Week 16, Grade 1 | 2 | 0 | 2 | 2
  Week 19, Grade 0: number analyzed (Participants) | 5 | 2 | 3 | 2
  Week 19, Grade 0 | 3 | 2 | 2 | 0
  Week 19, Grade 1: number analyzed (Participants) | 5 | 2 | 3 | 2
  Week 19, Grade 1 | 2 | 0 | 1 | 2
  Week 22, Grade 0: number analyzed (Participants) | 4 | 2 | 3 | 1
  Week 22, Grade 0 | 2 | 1 | 2 | 0
  Week 22, Grade 1: number analyzed (Participants) | 4 | 2 | 3 | 1
  Week 22, Grade 1 | 2 | 1 | 1 | 1
  Week 25, Grade 0: number analyzed (Participants) | 3 | 2 | 3 | 1
  Week 25, Grade 0 | 2 | 1 | 1 | 0
  Week 25, Grade 1: number analyzed (Participants) | 3 | 2 | 3 | 1
  Week 25, Grade 1 | 1 | 1 | 2 | 1
  Week 28, Grade 0: number analyzed (Participants) | 2 | 1 | 3 | 1
  Week 28, Grade 0 | 2 | 0 | 1 | 0
  Week 28, Grade 1: number analyzed (Participants) | 2 | 1 | 3 | 1
  Week 28, Grade 1 | 0 | 1 | 2 | 1
  Week 31, Grade 0: number analyzed (Participants) | 2 | 1 | 1 | 0
  Week 31, Grade 0 | 2 | 1 | 1 |
  Week 34, Grade 0: number analyzed (Participants) | 2 | 1 | 1 | 0
  Week 34, Grade 0 | 2 | 1 | 0 |
  Week 37, Grade 0: number analyzed (Participants) | 2 | 0 | 1 | 0
  Week 37, Grade 0 | 1 |  | 1 |
  Week 37, Grade 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Week 37, Grade 1 | 1 |  | 0 |
  Week 40, Grade 0: number analyzed (Participants) | 2 | 0 | 1 | 0
  Week 40, Grade 0 | 2 |  | 0 |
  Week 40, Grade 1: number analyzed (Participants) | 2 | 0 | 1 | 0
  Week 40, Grade 1 | 0 |  | 1 |
  Week 43, Grade 0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 43, Grade 0 | 1 |  | 0 |
  Week 43, Grade 1: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 43, Grade 1 | 0 |  | 1 |
  Week 46, Grade 0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 46, Grade 0 | 1 |  | 0 |
  Week 46, Grade 1: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 46, Grade 1 | 0 |  | 1 |
  Week 49, Grade 0: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 49, Grade 0 | 1 |  | 0 |
  Week 49, Grade 2: number analyzed (Participants) | 1 | 0 | 1 | 0
  Week 49, Grade 2 | 0 |  | 1 |
  Week 52, Grade 0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 52, Grade 0 | 1 |  |  |
  Week 55, Grade 0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 55, Grade 0 | 1 |  |  |
  Week 58, Grade 0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Week 58, Grade 0 | 1 |  |  |
  Treatment Discontinuation (up to 107 weeks), Grade 0: number analyzed (Participants) | 8 | 7 | 9 | 7
  Treatment Discontinuation (up to 107 weeks), Grade 0 | 1 | 1 | 4 | 1
  Treatment Discontinuation (up to 107 weeks), Grade 1: number analyzed (Participants) | 8 | 7 | 9 | 7
  Treatment Discontinuation (up to 107 weeks), Grade 1 | 5 | 6 | 4 | 5
  Treatment Discontinuation (up to 107 weeks), Grade 2: number analyzed (Participants) | 8 | 7 | 9 | 7
  Treatment Discontinuation (up to 107 weeks), Grade 2 | 1 | 0 | 1 | 1
  Treatment Discontinuation (up to 107 weeks), Grade 3: number analyzed (Participants) | 8 | 7 | 9 | 7
  Treatment Discontinuation (up to 107 weeks), Grade 3 | 1 | 0 | 0 | 0

8. Primary Outcome: Part 1: Number of Participants With Worst-case Post Baseline Increase From Baseline in Vital Signs (Arm 4)
Description: Vital signs including systolic blood pressure (SBP), diastolic BP (DBP), pulse rate (PR) and body temperature (BT) were measured for the participants. DBP: Grade 0 (<80 millimeters of mercury [mmHg]), Grade 1 (80-89 mmHg), Grade 2 (90-99 mmHg), Grade 3 (>=100 mmHg); SBP: Grade 0 (<120 mmHg), Grade 1 (120-139 mmHg), Grade 2 (140-159 mmHg), Grade 3 (>=160 mmHg); PR categories include: 'Decrease to < 60 beats per minutes [bpm]', 'Change to Normal' or 'No Change', and 'Increase to >100 bpm'; BT categories include 'Decrease to <=35 degrees Celsius °C', 'Change to Normal' or 'No Change', and 'Increase to >=38 °C'. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Worst Case Post-Baseline includes all scheduled and unscheduled visits post baseline.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 8
Participants
  Diastolic Blood Pressure, Any Grade Increase | 0 | 2 | 2
  Diastolic Blood Pressure, Increase to Grade 2 | 0 | 1 | 0
  Diastolic Blood Pressure, Increase to Grade 3 | 0 | 0 | 1
  Systolic Blood Pressure, Any Grade Increase | 1 | 2 | 3
  Systolic Blood Pressure, Increase to Grade 2 | 1 | 2 | 2
  Systolic Blood Pressure, Increase to Grade 3 | 0 | 0 | 1
  Heart Rate, Decrease to <60 bpm | 0 | 0 | 0
  Heart Rate, Change to Normal or No Change | 4 | 7 | 6
  Heart Rate, Increase to >100 bpm | 2 | 2 | 2
  Temperature, Decrease to <=35 °C | 0 | 0 | 0
  Temperature, Change to Normal or No Change | 6 | 9 | 6
  Temperature, Increase to >=38 °C | 0 | 0 | 2

9. Primary Outcome: Part 1: Number of Participants With Worst-case Post Baseline Increase From Baseline in Vital Signs (Arm 5)
Description: as for outcome 8
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 9
Participants
  Diastolic Blood Pressure, Any Grade Increase | 5 | 1 | 4 | 5
  Diastolic Blood Pressure, Increase to Grade 2 | 3 | 0 | 1 | 0
  Diastolic Blood Pressure, Increase to Grade 3 | 0 | 0 | 0 | 0
  Systolic Blood Pressure, Any Grade Increase | 4 | 2 | 5 | 4
  Systolic Blood Pressure, Increase to Grade 2 | 1 | 1 | 2 | 1
  Systolic Blood Pressure, Increase to Grade 3 | 1 | 0 | 0 | 2
  Heart Rate, Decrease to <60 bpm | 0 | 0 | 0 | 0
  Heart Rate, Change to Normal or No Change | 7 | 7 | 9 | 7
  Heart Rate, Increase to >100 bpm | 3 | 0 | 2 | 2
  Temperature, Decrease to <=35 C | 0 | 0 | 0 | 0
  Temperature, Change to Normal or No Change | 10 | 6 | 11 | 9
  Temperature, Increase to >=38 C | 0 | 1 | 0 | 0

10. Primary Outcome: Part 1: Number of Participants Who Received Concomitant Medications (Arm 4)
Description: Number of participants who received Concomitant medications is summarized.
Time Frame: Up to approximately 97 weeks
Population: Intent To Treat (ITT) population included all participants who were randomized to treatment regardless of whether the participants actually received study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 9
Participants | 6 | 9 | 9

11. Primary Outcome: Part 1: Number of Participants Who Received Concomitant Medications (Arm 5)
Description: Number of participants who received Concomitant medications is summarized.
Time Frame: Up to approximately 107 weeks
Population: Intent To Treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants | 10 | 7 | 11 | 10

12. Primary Outcome: Part 1: Number of Participants With Worst-case Post Baseline Relative to Baseline Electrocardiogram (ECG) Findings (Arm 4)
Description: Number of participants with worst-case post baseline (WCPB) from baseline ECG findings is summarized as clinically significant. Data is summarized as Normal, Abnormal - Not Clinically Significant (NCS) and Abnormal - Clinically Significant (CS). Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Worst Case Post-Baseline includes all scheduled and unscheduled visits post baseline.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 8 | 9
Participants
  Baseline: Normal | 4 | 2 | 4
  Baseline: Abnormal - NCS | 2 | 6 | 3
  Baseline: Abnormal - CS | 0 | 0 | 2
  Worst-case post baseline: number analyzed (Participants) | 5 | 4 | 8
  Worst-case post baseline: Normal | 2 | 2 | 3
  Worst-case post baseline: Abnormal - NCS | 3 | 1 | 2
  Worst-case post baseline: Abnormal - CS | 0 | 1 | 3

13. Primary Outcome: Part 1: Number of Participants With Worst-case Post Baseline Relative to Baseline ECG Findings (Arm 5)
Description: as for outcome 12
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants
  Baseline: Normal | 5 | 5 | 5 | 7
  Baseline: Abnormal - NCS | 4 | 1 | 5 | 2
  Baseline: Abnormal - CS | 1 | 1 | 1 | 1
  Worst-case post baseline: number analyzed (Participants) | 10 | 7 | 11 | 9
  Worst-case post baseline: Normal | 0 | 5 | 4 | 4
  Worst-case post baseline: Abnormal - NCS | 7 | 2 | 4 | 5
  Worst-case post baseline: Abnormal - CS | 3 | 0 | 3 | 0

14. Primary Outcome: Part 1: Number of Participants With Worst-case Post Baseline Relative to Baseline in QTcF Interval (Arm 4)
Description: The QTcF values based on Fridericia formula were rounded to the integer and the values are categorized into the following ranges, inclusively: Grade 0 (<450 millisecond (msec)), Grade 1 (≥450-≤480 msec), Grade 2 (≥481-≤500 msec), and Grade 3 (≥501 msec). Missing baseline grades were assumed to be Grade 0. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Worst Case Post-Baseline includes all scheduled and unscheduled visits post baseline.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 8 | 9
Participants
  Baseline, Grade 0 | 4 | 6 | 8
  Baseline, Grade 1 | 1 | 0 | 0
  Baseline, Grade 2 | 0 | 1 | 1
  Baseline, Grade 3 | 1 | 1 | 0
  WCPB, No Grade Increase: number analyzed (Participants) | 5 | 4 | 8
  WCPB, No Grade Increase | 4 | 4 | 7
  WCPB, Increase to Grade 1: number analyzed (Participants) | 5 | 4 | 8
  WCPB, Increase to Grade 1 | 1 | 0 | 1

15. Primary Outcome: Part 1: Number of Participants With Worst-case Post Baseline Relative to Baseline in QTcF Interval (Arm 5)
Description: as for outcome 14
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants
  Baseline, Grade 0: number analyzed (Participants) | 10 | 7 | 11 | 9
  Baseline, Grade 0 | 10 | 6 | 10 | 9
  Baseline, Grade 1: number analyzed (Participants) | 10 | 7 | 11 | 9
  Baseline, Grade 1 | 0 | 1 | 1 | 0
  Baseline, Grade 2: number analyzed (Participants) | 10 | 7 | 11 | 9
  Baseline, Grade 2 | 0 | 0 | 0 | 0
  Baseline, Grade 3: number analyzed (Participants) | 10 | 7 | 11 | 9
  Baseline, Grade 3 | 0 | 0 | 0 | 0
  WCPB, No Grade Increase: number analyzed (Participants) | 10 | 7 | 11 | 9
  WCPB, No Grade Increase | 10 | 5 | 11 | 8
  WCPB, Increase to Grade 2: number analyzed (Participants) | 10 | 7 | 11 | 9
  WCPB, Increase to Grade 2 | 0 | 2 | 0 | 0
  WCPB, Increase to Grade 3: number analyzed (Participants) | 10 | 7 | 11 | 9
  WCPB, Increase to Grade 3 | 0 | 0 | 0 | 1

16. Primary Outcome: Part 1: Number of Participants With Worst-case Post Baseline Relative to Baseline in Left Ventricular Ejection Fraction (LVEF) (Arm 4)
Description: Number of participants with worst case post-baseline in LVEF from baseline is summarized as 'any decrease (>0%-<10% Decrease, 10%-19% Decrease, >=20% Decrease)', '>=10% Decrease and >= Lower limit of normal (LLN)', '>=10% Decrease and < LLN', '>=20% Decrease and >= LLN' and '>=20% Decrease and < LLN' . An increase is defined as an increase in grade relative to Baseline grade. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Worst Case Post-Baseline includes all scheduled and unscheduled visits post baseline.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 0 | 1 | 0
Participants
  No change or any increase |  | 1 |
  Any Decrease |  | 0 |
  >=10% Decrease and >= LLN |  | 0 |
  >=10% Decrease and < LLN |  | 0 |
  >=20% Decrease and >= LLN |  | 0 |
  >=20% Decrease and < LLN |  | 0 |

17. Primary Outcome: Part 1: Number of Participants With Worst-case Post Baseline Relative to Baseline in Left Ventricular Ejection Fraction (LVEF) (Arm 5)
Description: as for outcome 16
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 2 | 0 | 2 | 1
Participants
  No change or any increase | 2 |  | 0 | 0
  Any Decrease | 0 |  | 2 | 1
  >=10% Decrease and >= LLN | 0 |  | 0 | 0
  >=10% Decrease and < LLN | 0 |  | 0 | 0
  >=20% Decrease and >= LLN | 0 |  | 0 | 0
  >=20% Decrease and < LLN | 0 |  | 0 | 0

18. Primary Outcome: Part 1: Number of Participants With Worst Case Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline (Arm 4)
Description: Blood samples were collected for the analysis of hematology parameters and are categorized in alignment with Common Terminology Criteria for Adverse Events (CTCAE) version 5 as Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; and Grade 4: life-threatening consequences. Higher grade indicates greater severity. An increase in grade is defined relative to the Baseline grade. Participants with missing baseline values are assumed to have baseline value of grade 0. Any worst-case post baseline increase in grade along with any increase to a maximum grade of 3 and 4 is summarized. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Worst Case Post-Baseline includes all scheduled and unscheduled visits post baseline.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 8
Participants
  Eosinophils, Any Grade Increase: number analyzed (Participants) | 5 | 9 | 8
  Eosinophils, Any Grade Increase | 1 | 2 | 0
  Eosinophils, Increase to Grade 3: number analyzed (Participants) | 5 | 9 | 8
  Eosinophils, Increase to Grade 3 | 0 | 0 | 0
  Eosinophils, Increase to Grade 4: number analyzed (Participants) | 5 | 9 | 8
  Eosinophils, Increase to Grade 4 | 0 | 0 | 0
  Lymphocyte count decreased, Any Grade Increase: number analyzed (Participants) | 5 | 9 | 8
  Lymphocyte count decreased, Any Grade Increase | 1 | 6 | 6
  Lymphocyte count decreased, Increase to Grade 3: number analyzed (Participants) | 5 | 9 | 8
  Lymphocyte count decreased, Increase to Grade 3 | 0 | 1 | 2
  Lymphocyte count decreased, Increase to Grade 4: number analyzed (Participants) | 5 | 9 | 8
  Lymphocyte count decreased, Increase to Grade 4 | 0 | 0 | 0
  Lymphocyte count increased, Any Grade Increase: number analyzed (Participants) | 5 | 9 | 8
  Lymphocyte count increased, Any Grade Increase | 0 | 0 | 0
  Lymphocyte count increased, Increase to Grade 3: number analyzed (Participants) | 5 | 9 | 8
  Lymphocyte count increased, Increase to Grade 3 | 0 | 0 | 0
  Lymphocyte count increased, Increase to Grade 4: number analyzed (Participants) | 5 | 9 | 8
  Lymphocyte count increased, Increase to Grade 4 | 0 | 0 | 0
  Platelet count decreased, Any Grade Increase | 0 | 1 | 0
  Platelet count decreased, Increase to Grade 3 | 0 | 0 | 0
  Platelet count decreased, Increase to Grade 4 | 0 | 0 | 0
  White blood cell decreased, Any Grade Increase | 0 | 1 | 2
  White blood cell decreased, Increase to Grade 3 | 0 | 0 | 0
  White blood cell decreased, Increase to Grade 4 | 0 | 0 | 0
  Anemia, Any Grade Increase | 4 | 3 | 1
  Anemia, Increase to Grade 3 | 0 | 1 | 0
  Anemia, Increase to Grade 4 | 0 | 0 | 0
  Hemoglobin increased, Any Grade Increase | 0 | 0 | 0
  Hemoglobin increased, Increase to Grade 3 | 0 | 0 | 0
  Hemoglobin increased, Increase to Grade 4 | 0 | 0 | 0
  Neutrophil count decreased, Any Grade Increase: number analyzed (Participants) | 5 | 9 | 8
  Neutrophil count decreased, Any Grade Increase | 0 | 0 | 0
  Neutrophil count decreased, Increase to Grade 3: number analyzed (Participants) | 5 | 9 | 8
  Neutrophil count decreased, Increase to Grade 3 | 0 | 0 | 0
  Neutrophil count decreased, Increase to Grade 4: number analyzed (Participants) | 5 | 9 | 8
  Neutrophil count decreased, Increase to Grade 4 | 0 | 0 | 0

19. Primary Outcome: Part 1: Number of Participants With Worst Case Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline (Arm 5)
Description: as for outcome 18
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants
  Eosinophils, Any Grade Increase: number analyzed (Participants) | 9 | 7 | 11 | 10
  Eosinophils, Any Grade Increase | 1 | 2 | 3 | 3
  Eosinophils, Increase to Grade 3: number analyzed (Participants) | 9 | 7 | 11 | 10
  Eosinophils, Increase to Grade 3 | 0 | 0 | 0 | 0
  Eosinophils, Increase to Grade 4: number analyzed (Participants) | 9 | 7 | 11 | 10
  Eosinophils, Increase to Grade 4 | 0 | 0 | 0 | 0
  Lymphocyte count decreased, Any Grade Increase: number analyzed (Participants) | 9 | 7 | 10 | 10
  Lymphocyte count decreased, Any Grade Increase | 8 | 4 | 8 | 8
  Lymphocyte count decreased, Increase to Grade 3: number analyzed (Participants) | 9 | 7 | 10 | 10
  Lymphocyte count decreased, Increase to Grade 3 | 3 | 1 | 4 | 3
  Lymphocyte count decreased, Increase to Grade 4: number analyzed (Participants) | 9 | 7 | 10 | 10
  Lymphocyte count decreased, Increase to Grade 4 | 1 | 0 | 1 | 0
  Lymphocyte count increased, Any Grade Increase: number analyzed (Participants) | 9 | 7 | 10 | 10
  Lymphocyte count increased, Any Grade Increase | 0 | 0 | 0 | 0
  Lymphocyte count increased, Increase to Grade 3: number analyzed (Participants) | 9 | 7 | 10 | 10
  Lymphocyte count increased, Increase to Grade 3 | 0 | 0 | 0 | 0
  Lymphocyte count increased, Increase to Grade 4: number analyzed (Participants) | 9 | 7 | 10 | 10
  Lymphocyte count increased, Increase to Grade 4 | 0 | 0 | 0 | 0
  Platelet count decreased, Any Grade Increase | 1 | 0 | 2 | 0
  Platelet count decreased, Increase to Grade 3 | 0 | 0 | 0 | 0
  Platelet count decreased, Increase to Grade 4 | 0 | 0 | 1 | 0
  White blood cell decreased, Any Grade Increase | 0 | 1 | 0 | 1
  White blood cell decreased, Increase to Grade 3 | 0 | 0 | 0 | 0
  White blood cell decreased, Increase to Grade 4 | 0 | 0 | 0 | 0
  Anemia, Any Grade Increase | 6 | 2 | 4 | 4
  Anemia, Increase to Grade 3 | 1 | 0 | 1 | 0
  Anemia, Increase to Grade 4 | 0 | 0 | 0 | 0
  Hemoglobin increased, Any Grade Increase | 2 | 0 | 0 | 0
  Hemoglobin increased, Increase to Grade 3 | 2 | 0 | 0 | 0
  Hemoglobin increased, Increase to Grade 4 | 0 | 0 | 0 | 0
  Neutrophil count decreased, Any Grade Increase | 0 | 1 | 1 | 0
  Neutrophil count decreased, Increase to Grade 3 | 0 | 0 | 1 | 0
  Neutrophil count decreased, Increase to Grade 4 | 0 | 0 | 0 | 0

20. Primary Outcome: Part 1: Number of Participants With Worst Case Clinical Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline (Arm 4)
Description: Blood samples were collected for the analysis of clinical chemistry parameters and are categorized in alignment with Common Terminology Criteria for Adverse Events (CTCAE) version 5 as Grade 1: mild; Grade 2: moderate; Grade 3: severe or medically significant; and Grade 4: life-threatening consequences. Higher grade indicates greater severity. An increase in grade is defined relative to the Baseline grade. Participants with missing baseline values are assumed to have baseline value of grade 0. Any worst-case post baseline increase in grade along with any increase to a maximum grade of 3 and 4 is summarized. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Worst Case Post-Baseline includes all scheduled and unscheduled visits post baseline.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 8
Participants
  Activated Partial Thromboplastin Time (aPTT), Any Grade Increase: number analyzed (Participants) | 0 | 0 | 0
  Activated Partial Thromboplastin Time (aPTT), Any Grade Increase | 0 | 0 | 0
  aPTT, Increase to Grade 3: number analyzed (Participants) | 0 | 0 | 0
  aPTT, Increase to Grade 3 | 0 | 0 | 0
  aPTT, Increase to Grade 4: number analyzed (Participants) | 0 | 0 | 0
  aPTT, Increase to Grade 4 | 0 | 0 | 0
  Glucose, Any Grade Increase | 0 | 2 | 0
  Glucose, Increase to Grade 3 | 0 | 0 | 0
  Glucose, Increase to Grade 4 | 0 | 0 | 0
  International normalized ratio (INR) increased, Any Grade Increase: number analyzed (Participants) | 0 | 0 | 0
  International normalized ratio (INR) increased, Any Grade Increase | 0 | 0 | 0
  INR increased, Increase to Grade 3: number analyzed (Participants) | 0 | 0 | 0
  INR increased, Increase to Grade 3 | 0 | 0 | 0
  INR increased, Increase to Grade 4: number analyzed (Participants) | 0 | 0 | 0
  INR increased, Increase to Grade 4 | 0 | 0 | 0
  Alkaline phosphatase (AP), Any Grade Increase | 1 | 3 | 1
  AP, Increase to Grade 3 | 0 | 0 | 0
  AP, Increase to Grade 4 | 0 | 0 | 0
  Alanine aminotransferase (ALT), Any Grade Increase: number analyzed (Participants) | 6 | 9 | 7
  Alanine aminotransferase (ALT), Any Grade Increase | 1 | 2 | 0
  ALT, Increase to Grade 3: number analyzed (Participants) | 6 | 9 | 7
  ALT, Increase to Grade 3 | 0 | 0 | 0
  ALT, Increase to Grade 4: number analyzed (Participants) | 6 | 9 | 7
  ALT, Increase to Grade 4 | 0 | 0 | 0
  Aspartate aminotransferase (AST), Any Grade Increase | 1 | 1 | 0
  AST, Increase to Grade 3 | 0 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0 | 0
  Bilirubin, Any Grade Increase | 0 | 1 | 0
  Bilirubin, Increase to Grade 3 | 0 | 0 | 0
  Bilirubin, Increase to Grade 4 | 0 | 0 | 0
  Creatinine, Any Grade Increase | 2 | 3 | 3
  Creatinine, Increase to Grade 3 | 0 | 0 | 0
  Creatinine, Increase to Grade 4 | 0 | 0 | 0
  Potassium, Any Grade Increase | 0 | 2 | 1
  Potassium, Increase to Grade 3 | 0 | 0 | 0
  Potassium, Increase to Grade 4 | 0 | 0 | 0
  Lactate Dehydrogenase, Any Grade Increase | 1 | 2 | 3
  Lactate Dehydrogenase, Increase to Grade 3 | 0 | 0 | 0
  Lactate Dehydrogenase, Increase to Grade 4 | 0 | 0 | 0
  Sodium, Any Grade Increase | 0 | 0 | 0
  Sodium, Increase to Grade 3 | 0 | 0 | 0
  Sodium, Increase to Grade 4 | 0 | 0 | 0
  Albumin, Any Grade Increase | 4 | 3 | 4
  Albumin, Increase to Grade 3 | 0 | 0 | 0
  Albumin, Increase to Grade 4 | 0 | 0 | 0

21. Primary Outcome: Part 1: Number of Participants With Worst Case Clinical Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline (Arm 5)
Description: as for outcome 20
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants
  aPTT, Any Grade Increase: number analyzed (Participants) | 0 | 0 | 0 | 0
  aPTT, Any Grade Increase | 0 | 0 | 0 | 0
  aPTT, Increase to Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  aPTT, Increase to Grade 3 | 0 | 0 | 0 | 0
  aPTT, Increase to Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0
  aPTT, Increase to Grade 4 | 0 | 0 | 0 | 0
  Glucose, Any Grade Increase: number analyzed (Participants) | 10 | 7 | 11 | 9
  Glucose, Any Grade Increase | 0 | 0 | 0 | 2
  Glucose, Increase to Grade 3: number analyzed (Participants) | 10 | 7 | 11 | 9
  Glucose, Increase to Grade 3 | 0 | 0 | 0 | 0
  Glucose, Increase to Grade 4: number analyzed (Participants) | 10 | 7 | 11 | 9
  Glucose, Increase to Grade 4 | 0 | 0 | 0 | 0
  INR increased, Any Grade Increase: number analyzed (Participants) | 0 | 0 | 0 | 0
  INR increased, Any Grade Increase | 0 | 0 | 0 | 0
  INR increased, Increase to Grade 3: number analyzed (Participants) | 0 | 0 | 0 | 0
  INR increased, Increase to Grade 3 | 0 | 0 | 0 | 0
  INR increased, Increase to Grade 4: number analyzed (Participants) | 0 | 0 | 0 | 0
  INR increased, Increase to Grade 4 | 0 | 0 | 0 | 0
  AP, Any Grade Increase | 3 | 1 | 1 | 2
  AP, Increase to Grade 3 | 0 | 0 | 0 | 0
  AP, Increase to Grade 4 | 0 | 0 | 0 | 0
  ALT, Any Grade Increase | 1 | 0 | 1 | 3
  ALT, Increase to Grade 3 | 0 | 0 | 0 | 1
  ALT, Increase to Grade 4 | 0 | 0 | 0 | 0
  AST, Any Grade Increase | 0 | 2 | 3 | 2
  AST, Increase to Grade 3 | 0 | 0 | 0 | 0
  AST, Increase to Grade 4 | 0 | 0 | 0 | 0
  Bilirubin, Any Grade Increase | 2 | 0 | 2 | 0
  Bilirubin, Increase to Grade 3 | 0 | 0 | 0 | 0
  Bilirubin, Increase to Grade 4 | 0 | 0 | 1 | 0
  Creatinine, Any Grade Increase | 3 | 3 | 3 | 4
  Creatinine, Increase to Grade 3 | 1 | 0 | 0 | 1
  Creatinine, Increase to Grade 4 | 0 | 0 | 0 | 0
  Potassium, Any Grade Increase | 1 | 0 | 2 | 2
  Potassium, Increase to Grade 3 | 0 | 0 | 0 | 0
  Potassium, Increase to Grade 4 | 0 | 0 | 0 | 0
  Lactate Dehydrogenase, Any Grade Increase | 2 | 0 | 4 | 4
  Lactate Dehydrogenase, Increase to Grade 3 | 0 | 0 | 0 | 0
  Lactate Dehydrogenase, Increase to Grade 4 | 0 | 0 | 0 | 0
  Sodium, Any Grade Increase | 0 | 0 | 0 | 0
  Sodium, Increase to Grade 3 | 0 | 0 | 0 | 0
  Sodium, Increase to Grade 4 | 0 | 0 | 0 | 0
  Albumin, Any Grade Increase | 6 | 4 | 4 | 1
  Albumin, Increase to Grade 3 | 0 | 1 | 0 | 0
  Albumin, Increase to Grade 4 | 0 | 0 | 0 | 0

22. Primary Outcome: Part 1: Number of Participants With Worst Case Change Post-baseline in Clinical Chemistry Parameters (Arm 4)
Description: Blood samples were collected for analysis of clinical chemistry. The summaries of worst-case post baseline (WCPB) from baseline (B) with respect to normal range was analyzed. Data is presented as "XXX B YYY, WCPB YYY", where XXX denotes lab parameter and YYY is high/normal/low. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Worst Case Post-Baseline includes all scheduled and unscheduled visits post baseline.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%.When lab values were not analyzed for some participants, the Number of Participants Analyzed will be less than the total across categories, allowing for a direct comparison without adding an "Unknown" or "Data missing" category.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 9
Participants
  Calcium, B High, WCPB High | 0 | 1 | 1
  Calcium, B High, WCPB Normal | 0 | 0 | 0
  Calcium, B High, WCPB Low | 0 | 0 | 0
  Calcium, B Normal, WCPB High | 2 | 0 | 1
  Calcium, B Normal, WCPB Normal | 4 | 0 | 5
  Calcium, B Normal, WCPB Low | 0 | 0 | 1
  Calcium, B Low, WCPB High | 0 | 2 | 0
  Calcium, B Low, WCPB Normal | 0 | 7 | 0
  Calcium, B Low, WCPB Low | 0 | 0 | 0
  Lipase, B High, WCPB High: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B High, WCPB High | 0 | 0 | 0
  Lipase, B High, WCPB Normal: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B High, WCPB Normal | 0 | 0 | 0
  Lipase, B High, WCPB Low: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B High, WCPB Low | 0 | 0 | 0
  Lipase, B Normal, WCPB High: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B Normal, WCPB High | 1 | 1 | 2
  Lipase, B Normal, WCPB Normal: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B Normal, WCPB Normal | 4 | 5 | 5
  Lipase, B Normal, WCPB Low: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B Normal, WCPB Low | 0 | 0 | 0
  Lipase, B Low, WCPB High: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B Low, WCPB High | 0 | 0 | 0
  Lipase, B Low, WCPB Normal: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B Low, WCPB Normal | 0 | 1 | 0
  Lipase, B Low, WCPB Low: number analyzed (Participants) | 5 | 7 | 7
  Lipase, B Low, WCPB Low | 0 | 0 | 0
  Amylase, B High, WCPB High: number analyzed (Participants) | 5 | 6 | 7
  Amylase, B High, WCPB High | 0 | 1 | 0
  Amylase, B High, WCPB Normal: number analyzed (Participants) | 5 | 6 | 7
  Amylase, B High, WCPB Normal | 0 | 0 | 0
  Amylase, B High, WCPB Low: number analyzed (Participants) | 5 | 6 | 7
  Amylase, B High, WCPB Low | 0 | 0 | 0
  Amylase, B Normal, WCPB High: number analyzed (Participants) | 5 | 6 | 7
  Amylase, B Normal, WCPB High | 0 | 0 | 1
  Amylase, B Normal, WCPB Normal: number analyzed (Participants) | 5 | 6 | 7
  Amylase, B Normal, WCPB Normal | 4 | 4 | 6
  Amylase, B Normal, WCPB Low: number analyzed (Participants) | 5 | 6 | 7
  Amylase, B Normal, WCPB Low | 1 | 1 | 0
  Amylase, B Low, WCPB High: number analyzed (Participants) | 5 | 6 | 7
  Amylase, B Low, WCPB High | 0 | 0 | 0
  Amylase, B Low, WCPB Normal: number analyzed (Participants) | 5 | 9 | 7
  Amylase, B Low, WCPB Normal | 0 | 0 | 0
  Amylase, B Low, WCPB Low: number analyzed (Participants) | 5 | 9 | 7
  Amylase, B Low, WCPB Low | 0 | 0 | 0
  Urea, B High, WCPB High: number analyzed (Participants) | 4 | 5 | 6
  Urea, B High, WCPB High | 0 | 2 | 0
  Urea, B High, WCPB Normal: number analyzed (Participants) | 4 | 5 | 6
  Urea, B High, WCPB Normal | 0 | 0 | 0
  Urea, B High, WCPB Low: number analyzed (Participants) | 4 | 5 | 6
  Urea, B High, WCPB Low | 0 | 0 | 0
  Urea, B Normal, WCPB High: number analyzed (Participants) | 4 | 5 | 6
  Urea, B Normal, WCPB High | 1 | 1 | 0
  Urea, B Normal, WCPB Normal: number analyzed (Participants) | 4 | 5 | 6
  Urea, B Normal, WCPB Normal | 1 | 1 | 5
  Urea, B Normal, WCPB Low: number analyzed (Participants) | 4 | 5 | 6
  Urea, B Normal, WCPB Low | 1 | 0 | 1
  Urea, B Low, WCPB High: number analyzed (Participants) | 4 | 5 | 6
  Urea, B Low, WCPB High | 0 | 0 | 0
  Urea, B Low, WCPB Normal: number analyzed (Participants) | 4 | 5 | 6
  Urea, B Low, WCPB Normal | 1 | 0 | 0
  Urea, B Low, WCPB Low: number analyzed (Participants) | 4 | 5 | 6
  Urea, B Low, WCPB Low | 0 | 1 | 0
  Free Triiodothyronine (T3), B High, WCPB High: number analyzed (Participants) | 2 | 4 | 6
  Free Triiodothyronine (T3), B High, WCPB High | 0 | 0 | 0
  T3, B High, WCPB Normal: number analyzed (Participants) | 2 | 4 | 6
  T3, B High, WCPB Normal | 0 | 0 | 0
  T3, B High, WCPB Low: number analyzed (Participants) | 2 | 4 | 6
  T3, B High, WCPB Low | 0 | 0 | 0
  T3, B Normal, WCPB High: number analyzed (Participants) | 2 | 4 | 6
  T3, B Normal, WCPB High | 0 | 0 | 1
  T3, B Normal, WCPB Normal: number analyzed (Participants) | 2 | 4 | 6
  T3, B Normal, WCPB Normal | 1 | 2 | 4
  T3, B Normal, WCPB Low: number analyzed (Participants) | 2 | 4 | 6
  T3, B Normal, WCPB Low | 1 | 2 | 1
  T3, B Low, WCPB High: number analyzed (Participants) | 2 | 4 | 6
  T3, B Low, WCPB High | 0 | 0 | 0
  T3, B Low, WCPB Normal: number analyzed (Participants) | 2 | 4 | 6
  T3, B Low, WCPB Normal | 0 | 0 | 0
  T3, B Low, WCPB Low: number analyzed (Participants) | 2 | 4 | 6
  T3, B Low, WCPB Low | 0 | 0 | 0
  Free Thyroxine (T4), B High, WCPB High: number analyzed (Participants) | 4 | 7 | 6
  Free Thyroxine (T4), B High, WCPB High | 0 | 0 | 0
  T4, B High, WCPB Normal: number analyzed (Participants) | 4 | 7 | 6
  T4, B High, WCPB Normal | 0 | 0 | 0
  T4, B High, WCPB Low: number analyzed (Participants) | 4 | 7 | 6
  T4, B High, WCPB Low | 0 | 0 | 0
  T4, B Normal, WCPB High: number analyzed (Participants) | 4 | 7 | 6
  T4, B Normal, WCPB High | 0 | 0 | 0
  T4, B Normal, WCPB Normal: number analyzed (Participants) | 4 | 7 | 6
  T4, B Normal, WCPB Normal | 4 | 6 | 5
  T4, B Normal, WCPB Low: number analyzed (Participants) | 4 | 7 | 6
  T4, B Normal, WCPB Low | 0 | 1 | 0
  T4, B Low, WCPB High: number analyzed (Participants) | 4 | 7 | 6
  T4, B Low, WCPB High | 0 | 0 | 1
  T4, B Low, WCPB Normal: number analyzed (Participants) | 4 | 7 | 6
  T4, B Low, WCPB Normal | 0 | 0 | 0
  T4, B Low, WCPB Low: number analyzed (Participants) | 4 | 7 | 6
  T4, B Low, WCPB Low | 0 | 0 | 0
  Troponin I, B High, WCPB High: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B High, WCPB High | 0 | 1 | 0
  Troponin I, B High, WCPB Normal: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B High, WCPB Normal | 0 | 0 | 0
  Troponin I, B High, WCPB Low: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B High, WCPB Low | 0 | 0 | 0
  Troponin I, B Normal, WCPB High: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B Normal, WCPB High | 0 | 2 | 0
  Troponin I, B Normal, WCPB Normal: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B Normal, WCPB Normal | 1 | 0 | 3
  Troponin I, B Normal, WCPB Low: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B Normal, WCPB Low | 0 | 0 | 0
  Troponin I, B Low, WCPB High: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B Low, WCPB High | 0 | 0 | 0
  Troponin I, B Low, WCPB Normal: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B Low, WCPB Normal | 0 | 0 | 0
  Troponin I, B Low, WCPB Low: number analyzed (Participants) | 1 | 3 | 3
  Troponin I, B Low, WCPB Low | 0 | 0 | 0
  Thyrotropin, B High, WCPB High: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B High, WCPB High | 1 | 0 | 0
  Thyrotropin, B High, WCPB Normal: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B High, WCPB Normal | 0 | 0 | 0
  Thyrotropin, B High, WCPB Low: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B High, WCPB Low | 0 | 0 | 0
  Thyrotropin, B Normal, WCPB High: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B Normal, WCPB High | 0 | 1 | 0
  Thyrotropin, B Normal, WCPB Normal: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B Normal, WCPB Normal | 3 | 4 | 2
  Thyrotropin, B Normal, WCPB Low: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B Normal, WCPB Low | 0 | 1 | 5
  Thyrotropin, B Low, WCPB High: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B Low, WCPB High | 0 | 0 | 0
  Thyrotropin, B Low, WCPB Normal: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B Low, WCPB Normal | 1 | 0 | 0
  Thyrotropin, B Low, WCPB Low: number analyzed (Participants) | 5 | 7 | 7
  Thyrotropin, B Low, WCPB Low | 0 | 0 | 0

23. Primary Outcome: Part 1: Number of Participants With Worst Case Change Post-baseline in Clinical Chemistry Parameters (Arm 5)
Description: as for outcome 22
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed. Participants were counted twice if the participants have values that changed 'To Low' and 'To High', so the percentages may not add to 100%. When lab values were not analyzed for some participants, the Number of Participants Analyzed will be less than the total across categories, allowing for a direct comparison without adding an "Unknown" or "Data missing" category.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Participants
  Calcium, B High, WCPB High | 0 | 0 | 0 | 0
  Calcium, B High, WCPB Normal | 0 | 0 | 0 | 1
  Calcium, B High, WCPB Low | 0 | 0 | 0 | 0
  Calcium, B Normal, WCPB High | 0 | 1 | 0 | 0
  Calcium, B Normal, WCPB Normal | 9 | 5 | 7 | 8
  Calcium, B Normal, WCPB Low | 1 | 1 | 3 | 1
  Calcium, B Low, WCPB High | 0 | 0 | 0 | 0
  Calcium, B Low, WCPB Normal | 0 | 0 | 1 | 0
  Calcium, B Low, WCPB Low | 0 | 0 | 0 | 0
  Lipase, B High, WCPB High: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B High, WCPB High | 2 | 0 | 0 | 0
  Lipase, B High, WCPB Normal: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B High, WCPB Normal | 0 | 0 | 0 | 0
  Lipase, B High, WCPB Low: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B High, WCPB Low | 0 | 0 | 0 | 0
  Lipase, B Normal, WCPB High: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B Normal, WCPB High | 0 | 1 | 2 | 3
  Lipase, B Normal, WCPB Normal: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B Normal, WCPB Normal | 5 | 2 | 6 | 6
  Lipase, B Normal, WCPB Low: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B Normal, WCPB Low | 0 | 0 | 1 | 0
  Lipase, B Low, WCPB High: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B Low, WCPB High | 0 | 0 | 0 | 0
  Lipase, B Low, WCPB Normal: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B Low, WCPB Normal | 0 | 0 | 0 | 0
  Lipase, B Low, WCPB Low: number analyzed (Participants) | 7 | 3 | 10 | 9
  Lipase, B Low, WCPB Low | 0 | 0 | 1 | 0
  Amylase, B High, WCPB High: number analyzed (Participants) | 7 | 3 | 10 | 9
  Amylase, B High, WCPB High | 1 | 1 | 1 | 1
  Amylase, B High, WCPB Normal: number analyzed (Participants) | 3 | 3 | 10 | 9
  Amylase, B High, WCPB Normal | 0 | 0 | 0 | 0
  Amylase, B High, WCPB Low: number analyzed (Participants) | 3 | 3 | 10 | 9
  Amylase, B High, WCPB Low | 0 | 0 | 0 | 0
  Amylase, B Normal, WCPB High: number analyzed (Participants) | 7 | 3 | 10 | 9
  Amylase, B Normal, WCPB High | 0 | 0 | 2 | 2
  Amylase, B Normal, WCPB Normal: number analyzed (Participants) | 7 | 3 | 10 | 9
  Amylase, B Normal, WCPB Normal | 6 | 1 | 7 | 6
  Amylase, B Normal, WCPB Low: number analyzed (Participants) | 7 | 3 | 10 | 9
  Amylase, B Normal, WCPB Low | 0 | 0 | 0 | 0
  Amylase, B Low, WCPB High: number analyzed (Participants) | 7 | 3 | 10 | 9
  Amylase, B Low, WCPB High | 0 | 0 | 0 | 0
  Amylase, B Low, WCPB Normal: number analyzed (Participants) | 7 | 3 | 10 | 9
  Amylase, B Low, WCPB Normal | 0 | 1 | 0 | 0
  Amylase, B Low, WCPB Low: number analyzed (Participants) | 7 | 3 | 10 | 9
  Amylase, B Low, WCPB Low | 0 | 0 | 0 | 0
  Urea, B High, WCPB High: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B High, WCPB High | 2 | 1 | 0 | 0
  Urea, B High, WCPB Normal: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B High, WCPB Normal | 0 | 0 | 0 | 0
  Urea, B High, WCPB Low: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B High, WCPB Low | 0 | 0 | 0 | 0
  Urea, B Normal, WCPB High: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B Normal, WCPB High | 1 | 1 | 2 | 4
  Urea, B Normal, WCPB Normal: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B Normal, WCPB Normal | 2 | 4 | 3 | 3
  Urea, B Normal, WCPB Low: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B Normal, WCPB Low | 1 | 0 | 1 | 1
  Urea, B Low, WCPB High: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B Low, WCPB High | 0 | 0 | 0 | 0
  Urea, B Low, WCPB Normal: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B Low, WCPB Normal | 0 | 0 | 0 | 0
  Urea, B Low, WCPB Low: number analyzed (Participants) | 6 | 6 | 6 | 8
  Urea, B Low, WCPB Low | 0 | 0 | 0 | 0
  Free Triiodothyronine (T3), B High, WCPB High: number analyzed (Participants) | 6 | 4 | 9 | 9
  Free Triiodothyronine (T3), B High, WCPB High | 0 | 0 | 1 | 0
  T3, B High, WCPB Normal: number analyzed (Participants) | 6 | 4 | 9 | 9
  T3, B High, WCPB Normal | 0 | 0 | 0 | 0
  T3, B High, WCPB Low: number analyzed (Participants) | 6 | 4 | 9 | 9
  T3, B High, WCPB Low | 0 | 0 | 0 | 0
  T3, B Normal, WCPB High: number analyzed (Participants) | 6 | 4 | 9 | 9
  T3, B Normal, WCPB High | 1 | 0 | 1 | 0
  T3, B Normal, WCPB Normal: number analyzed (Participants) | 6 | 4 | 9 | 9
  T3, B Normal, WCPB Normal | 3 | 3 | 6 | 8
  T3, B Normal, WCPB Low: number analyzed (Participants) | 6 | 4 | 9 | 9
  T3, B Normal, WCPB Low | 1 | 0 | 1 | 1
  T3, B Low, WCPB High: number analyzed (Participants) | 6 | 4 | 9 | 9
  T3, B Low, WCPB High | 0 | 0 | 0 | 0
  T3, B Low, WCPB Normal: number analyzed (Participants) | 6 | 4 | 9 | 9
  T3, B Low, WCPB Normal | 0 | 0 | 0 | 0
  T3, B Low, WCPB Low: number analyzed (Participants) | 6 | 4 | 9 | 9
  T3, B Low, WCPB Low | 2 | 1 | 0 | 0
  Free Thyroxine (T4), B High, WCPB High: number analyzed (Participants) | 8 | 4 | 9 | 9
  Free Thyroxine (T4), B High, WCPB High | 0 | 1 | 0 | 1
  T4, B High, WCPB Normal: number analyzed (Participants) | 8 | 4 | 9 | 9
  T4, B High, WCPB Normal | 0 | 0 | 0 | 0
  T4, B High, WCPB Low: number analyzed (Participants) | 8 | 4 | 9 | 9
  T4, B High, WCPB Low | 0 | 0 | 0 | 0
  T4, B Normal, WCPB High: number analyzed (Participants) | 8 | 4 | 9 | 9
  T4, B Normal, WCPB High | 0 | 0 | 1 | 0
  T4, B Normal, WCPB Normal: number analyzed (Participants) | 8 | 4 | 9 | 9
  T4, B Normal, WCPB Normal | 7 | 3 | 7 | 8
  T4, B Normal, WCPB Low: number analyzed (Participants) | 8 | 4 | 9 | 9
  T4, B Normal, WCPB Low | 1 | 0 | 1 | 0
  T4, B Low, WCPB High: number analyzed (Participants) | 8 | 4 | 9 | 9
  T4, B Low, WCPB High | 0 | 0 | 0 | 0
  T4, B Low, WCPB Normal: number analyzed (Participants) | 8 | 4 | 9 | 9
  T4, B Low, WCPB Normal | 0 | 0 | 0 | 0
  T4, B Low, WCPB Low: number analyzed (Participants) | 8 | 4 | 9 | 9
  T4, B Low, WCPB Low | 0 | 0 | 0 | 0
  Troponin I, B High, WCPB High: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B High, WCPB High | 0 | 0 | 0 | 0
  Troponin I, B High, WCPB Normal: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B High, WCPB Normal | 0 | 0 | 0 | 0
  Troponin I, B High, WCPB Low: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B High, WCPB Low | 0 | 0 | 0 | 0
  Troponin I, B Normal, WCPB High: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B Normal, WCPB High | 0 | 0 | 1 | 0
  Troponin I, B Normal, WCPB Normal: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B Normal, WCPB Normal | 2 | 1 | 5 | 6
  Troponin I, B Normal, WCPB Low: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B Normal, WCPB Low | 0 | 0 | 0 | 0
  Troponin I, B Low, WCPB High: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B Low, WCPB High | 0 | 0 | 0 | 0
  Troponin I, B Low, WCPB Normal: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B Low, WCPB Normal | 0 | 0 | 0 | 0
  Troponin I, B Low, WCPB Low: number analyzed (Participants) | 2 | 1 | 6 | 6
  Troponin I, B Low, WCPB Low | 0 | 0 | 0 | 0
  Thyrotropin, B High, WCPB High: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B High, WCPB High | 2 | 1 | 1 | 0
  Thyrotropin, B High, WCPB Normal: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B High, WCPB Normal | 0 | 0 | 0 | 1
  Thyrotropin, B High, WCPB Low: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B High, WCPB Low | 0 | 0 | 0 | 0
  Thyrotropin, B Normal, WCPB High: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B Normal, WCPB High | 2 | 1 | 1 | 0
  Thyrotropin, B Normal, WCPB Normal: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B Normal, WCPB Normal | 5 | 3 | 5 | 7
  Thyrotropin, B Normal, WCPB Low: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B Normal, WCPB Low | 0 | 0 | 2 | 1
  Thyrotropin, B Low, WCPB High: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B Low, WCPB High | 0 | 0 | 0 | 0
  Thyrotropin, B Low, WCPB Normal: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B Low, WCPB Normal | 0 | 0 | 1 | 0
  Thyrotropin, B Low, WCPB Low: number analyzed (Participants) | 9 | 5 | 9 | 9
  Thyrotropin, B Low, WCPB Low | 0 | 0 | 0 | 0

24. Primary Outcome: Part 1: Number of Participants With Worst-Case Urinalysis Results Post-Baseline Relative to Baseline (Arm 4)
Description: Urinalysis was performed. Participants with missing value at baseline are assumed to be negative at baseline. All increases are from baseline. Baseline is defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Up to approximately 97 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 5 | 7 | 8
Participants
  Occult Blood, No Change/Decreased | 4 | 6 | 7
  Occult Blood, Any Increase | 1 | 1 | 1
  Occult Blood, Unknown | 0 | 0 | 0
  Protein, No Change/Decreased | 3 | 2 | 7
  Protein, Any Increase | 2 | 4 | 1
  Protein, Unknown | 0 | 1 | 0

25. Primary Outcome: Part 1: Number of Participants With Worst-Case Urinalysis Results Post-Baseline Relative to Baseline (Arm 5)
Description: as for outcome 24
Time Frame: Up to approximately 107 weeks
Population: Safety Population. Only those participants with data available at specified parameters have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 6 | 11 | 8
Participants
  Occult Blood, No Change/Decreased | 4 | 5 | 6 | 6
  Occult Blood, Any Increase | 4 | 0 | 5 | 2
  Occult Blood, Unknown | 2 | 1 | 0 | 0
  Protein, No Change/Decreased: number analyzed (Participants) | 8 | 6 | 11 | 8
  Protein, No Change/Decreased | 3 | 5 | 5 | 7
  Protein, Any Increase: number analyzed (Participants) | 8 | 6 | 11 | 8
  Protein, Any Increase | 5 | 1 | 6 | 1
  Protein, Unknown: number analyzed (Participants) | 8 | 6 | 11 | 8
  Protein, Unknown | 0 | 0 | 0 | 0

26. Primary Outcome: Part 2: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to the date of death, irrespective of the cause of death.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Part 1: Objective Response Rate (ORR) (Arm 4)
Description: ORR is defined as the percentage of participants with a best overall confirmed Complete response (CR) or Partial response (PR) at any time as per disease-specific criteria per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete Response (CR) is defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline).
Time Frame: Up to approximately 97 weeks
Population: Intent To Treat (ITT) population.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 9
Percentage of Participants | 0 [0.0 to 45.9] | 0 [0.0 to 33.6] | 0 [0.0 to 33.6]

28. Secondary Outcome: Part 1: Objective Response Rate (ORR) (Arm 5)
Description: ORR is defined as the percentage of participants with a best overall confirmed CR or PR at any time as per disease-specific criteria per RECIST version 1.1. CR is defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline).
Time Frame: Up to approximately 107 weeks
Population: Intent To Treat (ITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Percentage of Participants | 0 [0.0 to 30.8] | 0 [0.0 to 41.0] | 9 [0.2 to 41.3] | 0 [0.0 to 30.8]

29. Secondary Outcome: Part 1: Disease Control Rate (DCR) (Arm 4)
Description: DCR is defined as the percentage of participants with a confirmed CR + PR at any time, plus SD =>12 weeks as per RECIST v1.1. Complete Response (CR) is defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: Up to approximately 97 weeks
Population: Intent To Treat (ITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 9
Percentage of Participants | 17 [0.4 to 64.1] | 22 [2.8 to 60.0] | 11 [0.3 to 48.2]

30. Secondary Outcome: Part 1: Disease Control Rate (DCR) (Arm 5)
Description: as for outcome 29
Time Frame: Up to approximately 107 weeks
Population: Intent To Treat (ITT) population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
Percentage of Participants | 40 [12.2 to 73.8] | 14 [0.4 to 57.9] | 27 [6.0 to 61.0] | 0 [0.0 to 30.8]

31. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) and Minimum Observed Concentration (Cmin) of Belrestotug (Arm 4)
Description: Blood samples were collected for pharmacokinetic analysis of Belrestotug.
Time Frame: Up to 21 days (Cycle 1)
Population: Pharmacokinetic (PK) population included all participants from the ITT Population from whom a blood sample is obtained and analyzed for PK concentration. PK parameters were only calculated for treatment cycles in which sufficient data were available to do so.
Measure: Mean (Standard Deviation); unit: Microgram/ millilitre (ug/mL)
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 8
Microgram/ millilitre (ug/mL)
  Cmax | 88.470 (92.2653) | 118.762 (46.4217) | 271.835 (77.5244)
  Cmin | 9.412 (5.6264) | 22.091 (8.4224) | 44.350 (24.4184)

32. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) and Minimum Observed Concentration (Cmin) of Belrestotug (Arm 5)
Description: Blood samples were collected for pharmacokinetic analysis of Belrestotug.
Time Frame: Up to 21 days (Cycle 1)
Population: Pharmacokinetic (PK) population. PK parameters were only calculated for treatment cycles in which sufficient data were available to do so.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 10 | 10
ug/mL
  Cmax | 126.386 (21.8676) | 137.837 (34.5390) | 153.377 (33.5154) | 22.967 (7.0701)
  Cmin | 19.408 (6.4103) | 20.752 (11.5836) | 153.069 (54.3450) | 21.693 (9.2699)

33. Secondary Outcome: Part 1: Cmax and Cmin of Dostarlimab (Arm 4)
Description: Blood samples were collected for pharmacokinetic analysis of Dostarlimab.
Time Frame: Up to 21 days (Cycle 1)
Population: Pharmacokinetic (PK) population. Only those participants with data available at specified time points have been analyzed. PK parameters were only calculated for treatment cycles in which sufficient data were available to do so.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]
Number analyzed (Participants) | 6 | 9 | 9
ug/mL
  Cmax: number analyzed (Participants) | 5 | 9 | 9
  Cmax | 119.400 (60.9173) | 124.278 (40.6026) | 97.433 (34.2035)
  Cmin: number analyzed (Participants) | 6 | 7 | 8
  Cmin | 33.900 (15.3454) | 34.071 (8.5638) | 22.935 (7.9792)

34. Secondary Outcome: Part 1: Cmax and Cmin of Dostarlimab (Arm 5)
Description: Blood samples were collected for pharmacokinetic analysis of Dostarlimab.
Time Frame: Up to 21 days (Cycle 1)
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 10 | 7 | 11 | 10
ug/mL
  Cmax | 108.920 (32.2323) | 126.857 (51.0830) | 68.751 (43.8090) | 109.330 (121.1920)
  Cmin: number analyzed (Participants) | 10 | 6 | 11 | 8
  Cmin | 29.290 (12.4519) | 34.550 (13.2960) | 34.218 (12.3900) | 39.013 (26.8319)

35. Secondary Outcome: Part 1: Cmax and Cmin of Nelistotug (Arm 5)
Description: Blood samples were collected for pharmacokinetic analysis of Nelistotug.
Time Frame: Up to 21 days (Cycle 1)
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 9 | 7 | 10 | 8
ug/mL
  Cmax | 299.889 (313.2561) | 479.714 (219.7148) | 75.580 (12.4318) | 554.750 (140.7792)
  Cmin | 43.689 (13.7240) | 88.243 (34.7201) | 15.070 (2.9601) | 123.975 (66.4588)

36. Secondary Outcome: Part 2: Survival Rate at 12 and 18 Months
Description: Survival rate was planned to be anaysed at 12 and 18 months
Time Frame: At 12 and 18 months
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

37. Secondary Outcome: Part 2: Number of Participants With Complete Response (CR), Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD)
Description: CR, PR, SD and PD was planned to be evaluated as per RECIST version 1.1 criteria. Complete Response (CR) is defined as disappearance of all target and non-target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease. Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

38. Secondary Outcome: Part 2: Progression-free Survival (PFS)
Description: PFS is defined as time from the date of randomization to the date of disease progression as per RECIST v1.1. or death whichever occurs earlier. Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

39. Secondary Outcome: Part 2: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a best overall confirmed Complete response (CR) or Partial response (PR) at any time as per disease-specific criteria per RECIST version 1.1. Complete Response (CR) is defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline).
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Part 2: Duration of Response (DOR)
Description: DOR is defined as the time for first documented evidence of CR or PR until disease progression or death, per RECIST 1.1 criteria. Complete Response (CR) is defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Part 2: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants with a confirmed CR + PR at any time, plus SD =>12 weeks as per RECIST v1.1. Complete Response (CR) is defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). Stable Disease (SD) is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Part 2: Number of Participants With Immune-based (i) Complete Response (iCR), Partial Response (iPR), Unconfirmed Progressive Disease (iUPD), Confirmed Progressive Disease (iCPD), and Stable Disease (iSD)
Description: Modified RECIST 1.1 for immune-based therapeutics (iRECIST) is based on RECIST v 1.1 but adapted to account for the unique tumor response seen with immunotherapeutic drugs. iRECIST is used to assess tumor response and progression and make treatment decisions. iCR: disappearance of all target lesions; iPR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters (e.g. percent change from baseline). iCPD: either 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; iSD: stable disease in the absence of CR or PD and iUPD: unconfirmed progressive disease when PD is unconfirmed and NE: not evaluable.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Part 2: Progression-free Survival (iPFS)
Description: iPFS is defined as time from the date of randomization to the date of disease progression or death, whichever occurs earlier, per iRECIST criteria. Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Part 2: Objective Response Rate (iORR)
Description: iORR is defined as the percentage of participants with a confirmed iCR or iPR at any time per iRECIST criteria. iCR is defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. iPR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Part 2: Duration of Response (iDOR)
Description: iDOR is defined as the time from first documented evidence of CR or PR until disease progression or death, per iRECIST criteria. iCR is defined as disappearance of all target and non target lesions and any pathological lymph nodes must be <10 millimeter (mm) in the short axis. iPR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference, the baseline sum of the diameters.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

46. Secondary Outcome: Part 2: Number of Participants With AEs, SAEs, Adverse Events of Special Interest (AESI), AE/SAEs Leading to Dose Modifications/Delays/Withdrawals
Description: An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect, any other situation such as important medical events according to medical or scientific judgement. AESI are considered to be Infusion Related Reactions (IRRs) and those of potential immunologic etiology. AEs were planned to be coded using the MedDRA coding system.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Part 2: Number of Participants With Clinically Significant Changes in Vital Signs and Laboratory Parameters
Description: Clinically significant changes in vital signs were planned to be assessed. Blood samples were planned to be collected for the analysis of laboratory parameters.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

48. Secondary Outcome: Part 2: Cmax and Cmin for Dostarlimab
Description: Blood samples were planned to be collected to assess the pharmacokinetics of Dostarlimab.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

49. Secondary Outcome: Part 2: Cmax and Cmin for Belrestotug
Description: Blood samples were planned to be collected to assess the pharmacokinetics of Belrestotug.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

50. Secondary Outcome: Part 2: Number of Participants With Positive Anti-drug Antibodies (ADA)
Description: Serum samples were planned to be collected for the analysis of the presence of ADAs using validated immunoassays.
Time Frame: Up to approximately 107 weeks
Population: No participants were enrolled in Part 2 of the study. Hence, data was not collected.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)] | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug HD
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-SAEs and SAEs were collected up to approximately 97 weeks for arm 4 and up to approximately 107 weeks for arm 5.
Description: Safety Population included all participants who received at least 1 dose of standard of care (SoC) or experimental regimen based on actual treatment received.
Groups:
- Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]): Participants with NSCLC were administered with 500 mg of Dostarlimab as IV infusion once Q3W in combination with Belrestotug HD as IV infusion Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met.
- Arm 5 Randomized Part: Belrestotug(MD) + Dostarlimab + Nelistotug (HD): Participants with NSCLC received 500 mg Dostarlimab followed by Belrestotug MD and Nelistotug HD. Treatment were given via IV infusion from day 1 to Q3W for maximum duration of approximately 2 years or up to 35 treatment visits whichever comes first, or until disease progression, death, unacceptable toxicity, or other protocol-defined criteria are met. In this randomization part, participants were assessed for PK/PD and received various dose levels.
Arm/Group | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]) | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD | Arm 5 Randomized Part: Belrestotug(MD) + Dostarlimab + Nelistotug (HD)
All-Cause Mortality (participants affected / at risk) | 4/6 | 5/9 | 7/9 | 7/10 | 4/7 | 7/11 | 6/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 3/9 | 2/9 | 3/10 | 3/7 | 3/11 | 3/10
Other Adverse Events (participants affected / at risk) | 6/6 | 9/9 | 8/9 | 10/10 | 6/7 | 11/11 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] (N=6) | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] (N=9) | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]) (N=9) | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD (N=10) | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD (N=7) | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD (N=11) | Arm 5 Randomized Part: Belrestotug(MD) + Dostarlimab + Nelistotug (HD) (N=10)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Strangulated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 4: Dostarlimab + Belrestotug [Low Dose (LD)] (N=6) | Arm 4: Dostarlimab + Belrestotug [Medium Dose (MD)] (N=9) | Arm 4: Dostarlimab + Belrestotug [High Dose (HD)]) (N=9) | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug MD (N=10) | Arm 5 Safety Part: Belrestotug MD + Dostarlimab + Nelistotug HD (N=7) | Arm 5 Randomized Part: Belrestotug MD + Dostarlimab + Nelistotug LD (N=11) | Arm 5 Randomized Part: Belrestotug(MD) + Dostarlimab + Nelistotug (HD) (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcapsular splenic haematoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 3 (3) | 2 (2)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Discomfort (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Contrast media allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (10) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Varicella zoster virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 5 (5) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood sodium increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cranial nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Azotaemia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Capillaritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (3) | 2 (2) | 2 (3) | 1 (2) | 2 (3) | 3 (5)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (3) | 2 (2) | 1 (1) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT06926673/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/73/NCT06926673/SAP_001.pdf